CLINICAL TRIAL: NCT02011282
Title: Electro-Neuro-Muscular Stimulation in Hospitalized Intensive Care Patients
Brief Title: Electro-Neuro-Muscular Stimulation in ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, DEMOSTHENES MAKRIS, ASS. Professor in Critical Care Medicine, University of Thessaly
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CIM-TRIAL
Record Dates: First submitted 2013-12-09; First posted 2013-12-13 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-08

CONDITIONS: Myopathy; Neuropathy
Keywords: ICU,; MYOPATHY,; NEUROPATHY,; PNEUMONIA
MeSH Terms: conditions — Muscular Diseases; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electro-Neuro-Muscular Stimulation (Experimental): Patients will receive daily sessions of electrostimulation with a commercially available device (En-Stimulation 4, Netherlands) in the quadriceps muscle for 10 days
  Interventions: Other: Patients will receive daily sessions of electro-neuro-stimulation in the quadriceps muscle for 10 days
- Control (No Intervention): Patients in this arm will receive the usual standard treatment

INTERVENTIONS:
Other: Patients will receive daily sessions of electro-neuro-stimulation in the quadriceps muscle for 10 days
  Arms: Electro-Neuro-Muscular Stimulation

SUMMARY:
We will examine whether the application of electro-neuro-muscular stimulation (ENMS) in critical care patients, can decrease the impact or severity of the critical illness myopathy (CIM) or neuropathy. We will also assess whether electro-neuro-muscular stimulation affect the incidence density rate of nosocomial pneumonia in the ICU.

Patients will be divided into two groups, Group A and Group B chosen at random. In Group A conventional physiotherapy will be applied while in Group B, ENMS will also be applied additional to physiotherapy, in the quadriceps muscles. The total time of applying ENMS will be 1 hour, it will be applied before the start of the physiotherapy per day of hospitalization and for 10 days in each patient.

The definition of CIM will be based on pathology muscular biopsy (quadriceps). Patients will undergo biopsy on the 1st and 11th day after entering the study. The technique of Gomori Trichrome will be used to determine the existence or absence of myopathy. In addition the ATPase technique will be applied at different prices of PH (PH: 9,4, PH: 4,6 and PH : 4.3), thus achieving a separation of myopathy and neuropathy.

The primary outcome of the study will be the incidence of myopathy in both groups, at day 12th. Considering that the incidence of myopathy in critically ill patients is 80% reducing this rate by 50% in the intervention group using statistical power equal to 0.80 up to a level of p <0.05, 12 number of patients will be required in each group.

ELIGIBILITY:
Inclusion Criteria:

Patients aged>18 years old and <85 years old, hospitalized in the ICU for at least 96 hours

Exclusion Criteria:

pregnancy, autoimmune disease, pre-existing known neuromuscular diseases, presence of bone fractures on the lower extremities, use of corticoids

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
incidence of myopathy | 12 days
  Presence of myopathy in critical care patients; myopathy will be assessed with biopsy of quadriceps at day 12 after entering the study (17 day of ICU hospitalization)

SECONDARY OUTCOMES:
NEUROPATHY | 12 days
  presence of peripheral neuropathy after 12 days of hospitalization in the ICU

OTHER OUTCOMES:
ventilator associated pneumonia | 28 days
  presence of ventilator associated pneumonia during 28 days of stay in the ICU

CONTACTS AND LOCATIONS:
Overall Officials: EPAMINONDAS ZAKYNTHINOS, PROF, Study Director — University of Thessaly
Locations (1):
- Icu University Hospital Larissa, Larissa, Thessaly, Greece